## STATISTICAL ANALYSIS PLAN

Descriptive statistics (mean, standard deviation) will be used to describe the participants involved and results of kinesiophobia cover scale, WOMAC scale, gait analysis and TUG. The spatiotemporal and kinetic parameters, electromyographic activation, TUG and postural control will be analyzed by analysis of variance 3x2 considering time factor (pre, post 6 weeks, post 6 months) and groups (with and without informative leaflet), respectively. If the sphericity hypothesis is rejected, the Huynh-Fedt correction will be applied. Effect sizes will be computed by means of partial square eta values. The SPSS 20.0 package will be used for all analyzes. The p value used will be 0.05.